CLINICAL TRIAL: NCT02976480
Title: The Irrigation or No Irrigation in Simple Lacerations Trials
Acronym: ION-SiLac
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Agence de la Sante et des Services Sociaux du Saguenay-Lac-Saint-Jean (Other)
Responsible Party: Principal Investigator, Julien Bouchard, MD, CCFP(EM), Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-025
Record Dates: First submitted 2016-11-03; First posted 2016-11-29 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Laceration - Injury; Infection
Keywords: Irrigation
MeSH Terms: conditions — Lacerations; Infections | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irrigation (Active Comparator): The subjects randomized to this group will have their simple lacerations irrigated with a normal saline solution.
  Interventions: Procedure: Irrigation
- No Irrigation (Experimental): The subjects randomized to this group will not have their simple lacerations directly irrigated with a normal saline solution.
  Interventions: Procedure: No irrigation

INTERVENTIONS:
Procedure: Irrigation — A designated unblinded medical team member (nurse, emergency room physician or resident/trainee uninvolved in that particular patient's care) will prepare the laceration for repair and perform the irrigation. Irrigation will be delivered through a 20 Gauge 1 inch long catheter mounted on a 60 millilitre syringe. The volume of normal saline used will be calculated as 60 millilitre per centimetre length of laceration for a maximum of 300 millilitre. Once completed, the treating physician will enter the room and proceed to the laceration closure with the method and equipment of his choice. Both the patient (through eye covering) and the treating physician will remain blinded to the intervention.
  Arms: Irrigation
Procedure: No irrigation — A designated unblinded medical team member (nurse, emergency room physician or resident/trainee uninvolved in that particular patient's care) will prepare the laceration for repair. The laceration will not directly be irrigated. In order to ensure blinding of the subjects, the surrounding of the wound will be irrigated with a total of 60 millilitre of normal saline delivered through a 20 Gauge 1 inch long catheter mounted on a 60 millilitre syringe. Care will be taken not to enter a margin of 5cm from the laceration edges. Once completed, the treating physician will enter the room and proceed to the laceration closure with the method and equipment of his choice. Both the patient (through eye covering) and the treating physician will remain blinded to the intervention.
  Arms: No Irrigation

SUMMARY:
The purpose of this study is to determine whether the irrigation or non-irrigation of a simple laceration treated in the emergency department has an effect on the subsequent rate of infection.

DETAILED DESCRIPTION:
Background: Current guidelines recommend that lacerations be irrigated prior to their closure. However, there is very little data in the literature suggesting that simple laceration irrigation diminishes the subsequent rate of infection. Do patients benefit from this practice that involves additional time and costs?

Hypothesis Testing & Procedure: The purpose of this double-blind randomized controlled non-inferiority study is to test the hypothesis that the non-irrigation of lacerations does not increase the rate of post-repair infection. Every adult patients presenting to the Chicoutimi's Hospital Emergency Department with a simple laceration will be identify by the triage nurse. Eligibility will subsequently be assessed by the emergency room physician according to the inclusion and exclusion criteria. Eligible and consenting patients will be randomized to either the irrigation or non-irrigation arm. Post-repair rate of infection and aesthetic appearance satisfaction will be reported.

Sample Size Determination: With the fairly liberal inclusion criteria, a 6% wound infection rate in the irrigation group is expected, which corresponds to the upper limit of the 2 to 6% range reported in the literature. Non-inferiority of non-irrigation would be accepted if the rate of infection in this group does not exceed by 4% the usual infection rate of 6% with irrigation, as previously stated. As such, for the study to be powered at 80% with a 95% one-sided confidence interval, a population of 874 patients would be needed to conclude that the non-irrigation is non-inferior when its infection rate does not exceed by more than 4% the infection rate of the irrigation group. In addition, to account for an attrition rate of approximately 10%, enrolment of 1000 patients is aimed.

Statistical Analysis: Statistical analysis will be done by a certified statistician. According to the distribution of our data, the Chi2 or the Fisher test will be used. A preliminary analysis of our data will be done in the Spring 2017 to assess safety of our intervention.

Plan for Missing Data: Patients that are lost at follow up will be considered as having had no infection if no record of subsequent visits for wound infection is found after consultation of the regional Electronic Medical Record.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* repair within 18 hours from time of injury
* repair done by the emergency room physician or trainee
* clean and simple lacerations (clean edge with no gross contamination, as assessed by the treating physician)

Exclusion Criteria:

* pregnant patients
* involving tendons, muscles, fascias, articulations
* located on the ear, nose or distal to metacarpophalangeal or metatarsophalangeal joint
* immunosuppressed (neutropenia, chronic corticotherapy, HIV, immunosuppressive therapy within 3 months)
* bite wounds
* lacerations with any loss of substance
* lacerations with foreign body
* complex lacerations (crush, stellate)
* grossly contaminated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
Laceration infection following repair | At 30 days post-repair
  The primary outcome measured will be the 30-day post-repair infection rate in both study groups.
  At 30 days post-repair, patients will be contacted by phone by a trained nurse. A standardized form will be used to collect relevant information. Patients will be asked whether they consulted a physician for a wound infection, and if antibiotics or drainage was required. An infected wound is defined as one requiring either drainage or antibiotic treatment by the assessing physician.
  The regional Medical Electronic Record will be reviewed for patients that were lost at follow up. Records of subsequent visits for wound infection will be looked for at 30 days post-repair.

SECONDARY OUTCOMES:
Laceration infections following repair | At 5 to 10 days post-repair
  The wounds of enrolled subjects will systematically be evaluated by a nurse between 5 to 10 days post-repair. A standardized form will be used by the nurse to identify criteria of possible wound infection (erythema, purulence, induration, fever, pain, fluctuance, dehiscence). A wound suspected to be infected by the presence of any of the previous criteria will immediately be evaluated by an emergency room physician to adjudicate on its infection status. An infected wound is defined as one requiring either drainage or antibiotic treatment based on the judgement of the physician.
  The regional Medical Electronic Record will be reviewed for patients that were lost at follow up. Records of subsequent visits for wound infection will be looked for at 30 days post-repair.
Aesthetic appearance of the laceration following repair | At 30 days post-repair
  The following question will be asked:
  "Considering the appearance and localisation of the laceration before repair, considering that complete healing of the laceration could take up to a year duration, and considering that sun exposure needs to be avoided during the healing period, are you satisfied with the appearance your laceration has today?" Yes or No.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Bouchard, MD, CCFP(EM), Principal Investigator — Université de Sherbrooke
Locations (1):
- CIUSSS Saguenay-Lac-St-Jean, Hôpital de Chicoutimi, Chicoutimi, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Dire DJ, Welsh AP. A comparison of wound irrigation solutions used in the emergency department. Ann Emerg Med. 1990 Jun;19(6):704-8. doi: 10.1016/s0196-0644(05)82484-9. PMID 2344089
- [Background] Moscati R, Mayrose J, Fincher L, Jehle D. Comparison of normal saline with tap water for wound irrigation. Am J Emerg Med. 1998 Jul;16(4):379-81. doi: 10.1016/s0735-6757(98)90133-4. PMID 9672456
- [Background] Moscati RM, Mayrose J, Reardon RF, Janicke DM, Jehle DV. A multicenter comparison of tap water versus sterile saline for wound irrigation. Acad Emerg Med. 2007 May;14(5):404-9. doi: 10.1197/j.aem.2007.01.007. PMID 17456554
- [Background] Griffiths RD, Fernandez RS, Ussia CA. Is tap water a safe alternative to normal saline for wound irrigation in the community setting? J Wound Care. 2001 Nov;10(10):407-11. doi: 10.12968/jowc.2001.10.10.26149. PMID 12964289
- [Background] Bansal BC, Wiebe RA, Perkins SD, Abramo TJ. Tap water for irrigation of lacerations. Am J Emerg Med. 2002 Sep;20(5):469-72. doi: 10.1053/ajem.2002.35501. PMID 12216046
- [Background] Valente JH, Forti RJ, Freundlich LF, Zandieh SO, Crain EF. Wound irrigation in children: saline solution or tap water? Ann Emerg Med. 2003 May;41(5):609-16. doi: 10.1067/mem.2003.137. PMID 12712026
- [Background] Fernandez R, Griffiths R. Water for wound cleansing. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD003861. doi: 10.1002/14651858.CD003861.pub3. PMID 22336796
- [Background] Stevenson TR, Thacker JG, Rodeheaver GT, Bacchetta C, Edgerton MT, Edlich RF. Cleansing the traumatic wound by high pressure syringe irrigation. JACEP. 1976 Jan;5(1):17-21. doi: 10.1016/s0361-1124(76)80160-8. PMID 933383
- [Background] Hollander JE, Richman PB, Werblud M, Miller T, Huggler J, Singer AJ. Irrigation in facial and scalp lacerations: does it alter outcome? Ann Emerg Med. 1998 Jan;31(1):73-7. doi: 10.1016/s0196-0644(98)70284-7. PMID 9437345
- [Background] Hollander JE, Singer AJ, Valentine S. Comparison of wound care practices in pediatric and adult lacerations repaired in the emergency department. Pediatr Emerg Care. 1998 Feb;14(1):15-8. doi: 10.1097/00006565-199802000-00004. PMID 9516624
- [Background] Maharaj D, Sharma D, Ramdass M, Naraynsingh V. Closure of traumatic wounds without cleaning and suturing. Postgrad Med J. 2002 May;78(919):281-2. doi: 10.1136/pmj.78.919.281. PMID 12151570
- [Background] Webster DJ, Davis PW. Closure of abdominal wounds by adhesive strips: a clinical trial. Br Med J. 1975 Sep 20;3(5985):696-8. doi: 10.1136/bmj.3.5985.696. PMID 1100188
- [Background] Rodeheaver GT, Pettry D, Thacker JG, Edgerton MT, Edlich RF. Wound cleansing by high pressure irrigation. Surg Gynecol Obstet. 1975 Sep;141(3):357-62. PMID 808870
- [Background] Longmire AW, Broom LA, Burch J. Wound infection following high-pressure syringe and needle irrigation. Am J Emerg Med. 1987 Mar;5(2):179-81. doi: 10.1016/0735-6757(87)90121-5. No abstract available. PMID 3828025
- [Background] Pronchik D, Barber C, Rittenhouse S. Low- versus high-pressure irrigation techniques in Staphylococcus aureus-inoculated wounds. Am J Emerg Med. 1999 Mar;17(2):121-4. doi: 10.1016/s0735-6757(99)90041-4. PMID 10102307
- [Background] Singer AJ, Hollander JE, Quinn JV. Evaluation and management of traumatic lacerations. N Engl J Med. 1997 Oct 16;337(16):1142-8. doi: 10.1056/NEJM199710163371607. No abstract available. PMID 9329936
- [Background] Hollander JE, Singer AJ. Laceration management. Ann Emerg Med. 1999 Sep;34(3):356-67. doi: 10.1016/s0196-0644(99)70131-9. PMID 10459093
- [Background] Nicks BA, Ayello EA, Woo K, Nitzki-George D, Sibbald RG. Acute wound management: revisiting the approach to assessment, irrigation, and closure considerations. Int J Emerg Med. 2010 Aug 27;3(4):399-407. doi: 10.1007/s12245-010-0217-5. PMID 21373312